CLINICAL TRIAL: NCT06089239
Title: De-Implementing Fall Prevention Alarms in Hospitals
Brief Title: Choosing Wisely: De-implementing Fall Prevention Alarms in Hospitals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CED000000718; R01AG073408-01A1 (NIH)
Record Dates: First submitted 2023-09-18; First posted 2023-10-18 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Accidental Fall; Patient Safety; Hospital Acquired Condition; Clinical Alarms; Mentoring
MeSH Terms: conditions — Iatrogenic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Coaching (Active Comparator): In Quarter 1, high intensity initiation coaching will consist of a four-hour orientation session that will include:
  * comprehensive information on behavior and organizational change theory,
  * suggested approaches, and
  * in-depth training on behavioral and organization-focused change techniques to stimulate implementation efforts.
  Commencing in Quarter 2, high intensity sustainability coaching will consist of:
  * weekly virtual follow up sessions for the first month, followed by private monthly coaching follow up sessions via a virtual format.
  * Access to additional monthly web-based, synchronous "office hours" for group discussion on progress and customized troubleshooting to assist in navigating barriers.
  * Sites will also have access to "on call" assistance with coaches to assist with navigating challenges in real time.
  Interventions: Other: High Intensity Coaching
- Low Intensity Coaching (Sham Comparator): In Quarter 1, low intensity initiation coaching will be conducted. It will consist of:
  * initial two-hour orientation session with introductory content on behavior change and organizational change theory and techniques,
  * an overview of implementation phases, and
  * selection of tailored de-implementation strategies for that site based on readiness for change, focus group data and local resources.
  Implementation coaches will provide the Fuld Toolkit for the site with suggestions for assigning strategies, local leaders, and development of timelines for de-implementation.
  Coaches will instruct site Team Leaders to establish the primary mechanism for sharing baseline and trended data in real time.
  Interventions: Other: Low Intensity Coaching

INTERVENTIONS:
Other: High Intensity Coaching — External coaching is a commonly used strategy to change practice, especially for multi-site collaboratives where implementation requires customization to the site. Coaches serve as skill builders who train organizational personnel in quality improvement processes and develop proficiency in the targeted practice area (i.e., fall prevention).
  Arms: High Intensity Coaching
Other: Low Intensity Coaching — External coaching is a commonly used strategy to change practice, especially for multi-site collaboratives where implementation requires customization to the site. Coaches serve as skill builders who train organizational personnel in quality improvement processes and develop proficiency in the targeted practice area (i.e., fall prevention).
  Arms: Low Intensity Coaching

SUMMARY:
This is a Hybrid II de-implementation study to reduce use of fall prevention alarms in hospitals. The intervention consists of tailored, site-specific approaches for three core implementation strategies: education, audit/feedback and opinion leaders. Hospital units will be randomized to low-intensity or high-intensity coaching for the implementation of the tailored strategies.

DETAILED DESCRIPTION:
Inpatient falls result in significant physical and economic burdens to patients (increased injury and mortality rates and decreased quality of life) as well as to medical organizations (increased lengths of stay, medical care costs, and litigation). The Centers for Medicare & Medicaid Services (CMS) considers falls with injury a "never event"- an error in medical care that indicates a real problem in the safety and credibility of a health care institution. Hospitals are no longer reimbursed for extra costs incurred in the diagnosis and management of inpatient fall-related injuries. Thus, because patient falls are common, costly and interpreted as poor care quality, hospitals are highly incentivized to prevent them.

Alarm systems are designed to reduce falls by alerting staff when patients attempt to leave a bed or chair without assistance. There is now strong evidence that alarms are ineffective as a fall prevention maneuver in hospitals. Despite this, more than one-third of hospital patients are undergoing fall prevention alarm monitoring. In nursing homes, CMS regulates the use of fall prevention alarms as it does physical restraints. Instructions to nursing home surveyors state these devices should be used only when medically necessary and continuously reevaluated.

Guided by the Choosing Wisely De-implementation Framework, this project will generate a generalizable approach using coaching and tailored de-implementation strategies to reduce use of fall prevention alarms in hospitals. The investigators will conduct a hybrid II implementation study in 30 medical or medical-surgical units from US non-federal hospitals participating in the National Database of Nursing Quality Indicators. Findings from this study could also support future trials aimed at de-implementing low-quality alarm use in other care settings with known high fall rates (e.g., stroke care, cancer care). Evaluation of high versus low intensity coaching addresses an urgent need to evaluate use of tailored strategies and to establish effective thresholds for coaching within health service settings that have varying resources to support de-implementation efforts

ELIGIBILITY:
Inclusion Criteria:

* Stakeholders in fall prevention at up to 30 participating NDNQI hospitals

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Fall Prevention Alarm Prevalence survey | monthly for 30 months
  Number of Patients in a study unit with fall prevention alarm activated divided by the number of patients evaluated. This is assessed monthly and is expressed as the proportion of patients assessed with fall prevention alarm activated. This is not a time to event outcome.
  This measure will be recorded monthly for 30 months during both baseline and intervention periods.
Patient Falls | monthly for 30 months
  Patients on participating units are monitored for falls beginning the date/time they are admitted to the date/time they are discharged from the study unit. Falls are determined using National Database of Nursing Quality Indicators (NDNQI) protocols. Patients may contribute one or more falls during their stay. This is expressed as the Number of Patients who fell/1000 bed days of care.
  This measure will be recorded monthly for 30 months during both baseline and intervention periods.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald I Shorr, MD, Principal Investigator — University of Florida
Locations (24):
- United States (24):
  - PIH Health Downey Hospital, Downey, California
  - El Camino Health - Los Gatos, Mountain View, California
  - University of California Davis Medical Center, Sacramento, California
  - Lakeland Regional Medical Center, Lakeland, Florida
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - Hendricks Regional Health, Danville, Indiana
  - IU Health North Hospital, Indianapolis, Indiana
  - UMass Memorial Health Harrington, Southbridge, Massachusetts
  - Henry Ford Hospital West Bloomfield, West Bloomfield, Michigan
  - Lahey Hospital & Medical Center, Derry, New Hampshire
  - Hunterdon Medical Center, Flemington, New Jersey
  - Raritan Bay Medical Center, New Brunswick, New Jersey
  - Greenwich Hospital, River Vale, New Jersey
  - St Peter's Health Samaritan Hospital, Albany, New York
  - Grant Medical Center, Columbus, Ohio
  - Barberton Hospital, Uniontown, Ohio
  - Kaiser Westside Medical Center, Hillsboro, Oregon
  - Kaiser Permanente - Sunnyside Medical Center, Woodburn, Oregon
  - Christiana Care, West Chester, Pennsylvania
  - Kent Hospital, Warwick, Rhode Island
  - Prisma Health, Irmo, South Carolina
  - St. David's Medical Center, Austin, Texas
  - Covenant Medical Center, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turner K, McNett M, Potter C, Cramer E, Al Taweel M, Shorr RI, Mion LC. Alarm with care-a de-implementation strategy to reduce fall prevention alarm use in US hospitals: a study protocol for a hybrid 2 effectiveness-implementation trial. Implement Sci. 2023 Dec 5;18(1):70. doi: 10.1186/s13012-023-01325-9. PMID 38053114